CLINICAL TRIAL: NCT01407887
Title: Efficacy and Safety of Artesunate-amodiaquine Combined With Methylene Blue for Falciparum Malaria Treatment in African Children
Brief Title: Efficacy and Safety of Artesunate-amodiaquine-methylene for Malaria Treatment in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Olaf Müller, Prof Dr, Institut of Public Health, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFB544A8
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2011-06

CONDITIONS: Uncomplicated Falciparum Malaria
Keywords: children
MeSH Terms: interventions — Artesunate; Amodiaquine; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- artesunate, amodiaquine methylene blue (Active Comparator): two arms, open randomized controlled study in children with uncomplicated falciparum malaria in Burkina Faso. Intervention: artesunate (AS) - amodiaquine (AQ) - methylene blue (MB) control: artesunate (AS) - amodiaquine (AQ)
  Interventions: Drug: artesunate (AS) - amodiaquine (AQ) - methylene blue (MB)
- artesunate amodiaquine (No Intervention): The control group will receive once daily a fixed dose AS-AQ over three days.

INTERVENTIONS:
Drug: artesunate (AS) - amodiaquine (AQ) - methylene blue (MB) — The group AS-AQ-MB will receive once daily a fixed dose AS-AQ formulation combined with once daily MB over a three days period.
  Arms: artesunate, amodiaquine methylene blue

SUMMARY:
Title: Efficacy and safety of artesunate-amodiaquine combined with methylene blue for falciparum malaria treatment in African children: randomised controlled trial.

Design: Mono-centre, two arms, open randomized controlled study in children with uncomplicated falciparum malaria in Burkina Faso.

Phase: Phase II.

Objectives: The primary objective of this trial is to study the efficacy and safety of the triple therapy artesunate (AS) - amodiaquine (AQ) - methylene blue (MB) given over three days in young children with uncomplicated falciparum malaria in Burkina Faso compared to the local standard three days artemisinin-based combination therapy (ACT) AS-AQ regimen.

Population: Children aged 6-59 months with uncomplicated falciparum malaria from Nouna Hospital in north-western Burkina Faso.

Sample size: 180 patients (90 per study arm).

ELIGIBILITY:
Inclusion Criteria:

* 6-59 months old children (male and female)
* Weight ≥ 6kg
* Uncomplicated malaria caused by P. falciparum
* Asexual parasites ≥ 2 000/µl and ≤ 200 000/µl
* Axillary temperature ≥ 37.5°C or a history of fever during last 24 hours
* Burkinabe nationality
* Permanent residence in the study area with no intention of leaving during the surveillance period
* Informed consent

Exclusion Criteria:

* Severe malaria (WHO 2000)
* Vomiting (3 or more within 24 hours before the visit)
* Any apparent significant disease, including severe malnutrition
* A history of a previous, significant adverse reaction to either of the study drugs
* Anaemia (haemoglobin < 7 g/dl)
* Treated in the same trial before
* All modern antimalarial treatment prior to inclusion (last seven days)
* Simultaneous participation in another investigational study
* Treatment with other investigational drugs

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
P. falciparum gametocyte prevalence | day 14 of follow-up
  P. falciparum gametocyte prevalence on day 14 of follow-up (PCR determination)

SECONDARY OUTCOMES:
P. falciparum gametocyte prevalence and density | day 1, 2, 3, 7, and 28 of follow-up
  P. falciparum gametocyte prevalence and density on day 1, 2, 3, 7, and 28 of follow-up (PCR determination) P. falciparum gametocyte prevalence and density on day 1, 2, 3, 7, and 28 of follow-up (microscopic determination)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Müller, Prof Dr, Principal Investigator — Institut of Public health, University of heidelberg
Locations (1):
- Nouna Health District, Nouna, Mouhoun, Burkina Faso

REFERENCES:
- [Derived] Coulibaly B, Pritsch M, Bountogo M, Meissner PE, Nebie E, Klose C, Kieser M, Berens-Riha N, Wieser A, Sirima SB, Breitkreutz J, Schirmer RH, Sie A, Mockenhaupt FP, Drakeley C, Bousema T, Muller O. Efficacy and safety of triple combination therapy with artesunate-amodiaquine-methylene blue for falciparum malaria in children: a randomized controlled trial in Burkina Faso. J Infect Dis. 2015 Mar 1;211(5):689-97. doi: 10.1093/infdis/jiu540. Epub 2014 Sep 28. PMID 25267980